CLINICAL TRIAL: NCT04181840
Title: Impedance Spectroscopy Using the ONIRY Device in the Diagnosis of Sphincter Injuries in Women After Vaginal Deliveries
Brief Title: Impedance Spectroscopy for Obstetric Anal Sphincter Injuries Detection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OASIS Diagnostics S.A. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2/1/2019 (May 6)
Record Dates: First submitted 2019-11-21; First posted 2019-12-02 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Obstetric Anal Sphincter Injury; Delivery Complication; Obstetric Complication
Keywords: Obstetric Anal Sphincter Injury; Impedance Spectroscopy
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Impedance spectroscopy (Experimental): Maximum 56 women up to 16 weeks from a natural delivery, with at least one perinatal anal sphincter injury risk factor, such as: the extended second delivery phase, instrumental delivery (vacuum or forceps), shoulder dystocia, birth weight of the child > 4kg, episiotomy, uncontrolled perineal laceration (in patients with crotch protection).
  The planned interventions are:
  * Blood and faeces tests
  * Impedance spectroscopy test
  * Full gynecological and proctological examination
  * Transanal ultrasonography
  * Anorectal manometry
  Interventions: Diagnostic Test: Blood and faeces tests; Device: Impedance spectroscopy test; Diagnostic Test: Full gynecological and proctological examination; Diagnostic Test: Transanal ultrasonography; Diagnostic Test: Anorectal manometry; Other: Determining the degree of sphincter injury

INTERVENTIONS:
Diagnostic Test: Blood and faeces tests — During V1 - Laboratory tests, particularly for calprotectin concentration assessment
Device: Impedance spectroscopy test — During V1 - the electrical impedance of anal sphincter muscles will be measured
Diagnostic Test: Full gynecological and proctological examination — During V1 and V2 - Examination with a gynecological speculum, Two-handed examination, Rectal examination, and Anoscopy
Diagnostic Test: Transanal ultrasonography — During V1 - reference diagnostic methods with documented effectiveness and safety; for comparison with impedance spectroscopy results.
Diagnostic Test: Anorectal manometry — During V1 - reference diagnostic methods with documented effectiveness and safety; for comparison with impedance spectroscopy results.
Other: Determining the degree of sphincter injury — During V2 - conducting the examination will finally determine the extent of sphincter damage, present the patient with therapeutic options and decide on the treatment or rehabilitation of sphincter.

SUMMARY:
The main purpose of the study is to evaluate the effectiveness and safety of the impedance spectroscopy device prototype in the detection of anal sphincter injuries in women in the early postpartum period. The study is prospective. The study group comprises up to 56 patients; up to 16 weeks from a natural delivery. The planned participation of each patient in the study is up to 4 weeks and two visits will take place at that time.

After obtaining written consent, at the first visit (V1) each patient will undergo a physical examination (both proctological and gynecological examination), blood samples for laboratory tests and stool samples for calprotectin concentration assessment will be collected. The presence of clinical symptoms of both gas and stool incontinence will be assessed during the visit with the use of Wexner's scale. Then, the dates of two reference tests will be planned: Trans-rectal USG and Recto-anal manometry which will be performed as part of the V1 visit within a period not exceeding 27 days.

The V2 visit, which will also be the final visit, will include a reassessment of the patient's general condition, recording the values of basic vital parameters, subjective and physical examination, and then the doctor conducting the examination will finally determine the extent of sphincter damage, present the patient with therapeutic options and decide on the treatment or rehabilitation of sphincter.

During the visits, all adverse events will also be monitored, both those reported by patients and those related to the examined diagnostic device.

ELIGIBILITY:
Inclusion Criteria:

* women patients,
* 18-49 years old,
* up to 16 weeks from a natural delivery
* with the presence of:

  1. clinically confirmed OASIS at least stage II, as a result of an episiotomy or uncontrolled crotch rupture (in patients with crotch protection), or
  2. at least one risk factor, such as:
* the extended second delivery phase,
* instrumental delivery (vacuum or forceps),
* shoulder dystocia,
* birth weight of the child > 4kg,
* episiotomy,
* uncontrolled perineal laceration (in patients with crotch protection),
* induction of delivery using oxytocin,
* head circumference ≥34 mm and other.
* the patient's understanding of the nature of the clinical study and permission in writing from the patient to participate in this study.

Exclusion Criteria:

* the presence of acute diseases during treatment,
* the presence of chronic diseases not treated or treated insufficiently (e.g., incorrectly controlled hypertension),
* the presence of diseases with accompanying symptoms of fecal incontinence history of proctology surgery's whit postoperative complication,
* the presence of inflammatory bowel diseases during the exacerbation phase,
* the treatment in the last year because of serious, progressive, uncontrolled cardiological, pulmonary, nephrology, contagious or psychiatric illness whose course could affect the patient's risk increase due to participation in the study,
* significant disease symptoms so far undiagnosed,
* the presence or suspected malignant disease or previous on previous oncological treatment in the last 5 years,
* the presence of a cardiac stimulator or cardioverter-defibrillator,
* severe surgery or severe trauma in the last year.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-06-26 (Actual); Study Completion 2020-07-20 (Actual)

PRIMARY OUTCOMES:
Anal sphincters continuity (injuries) assessed in physical examination and trancanal ultrasonography | 16 weeks
  Assessment using:
  1. OASIS classification of perineal tears.
  2. Starck scale (0-16 scale, no defect - 0, maximum - 16, which means severe damage of both sphincters on a considerable length and circumference).
  3. Norderval scale (0-7 scale, no defect - 0, 7 is the maximal damage of both anal sphincters).
Anal sphincter tension (function) assessed in physical examination and anorectal manometry | 16 weeks
Anal sphincter assessment evaluated by impedance spectroscopy | 16 weeks
  Estimation of the presence, extent and severity of anal sphincter injury, by impedance moduli and phase shifts.
  The main aim of the study is to establish whether the extension and severity of obstetric anal sphincter injury can be precisely assessed with parameters calculated from anal sphincter muscles using impedance spectroscopy.

SECONDARY OUTCOMES:
Adverse events | 16 weeks
  Evaluation of the frequency and intensity of adverse events associated with the use of the new diagnostic method.

CONTACTS AND LOCATIONS:
Overall Officials: Małgorzata Uchman-Musielak, MD, PhD, Principal Investigator — Specialist Medical Practice
Locations (1):
- Praktyka Lekarska Małgorzata Uchman-Musielak, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor's website — http://www.oasis-diagnostics.eu